CLINICAL TRIAL: NCT02031796
Title: Cardiac Vascular Reconstruction (CAVAREC) DynaCT for 3D Assessment of Aortic Valve During TAVI Procedures
Brief Title: Cardiac Vascular Reconstruction DynaCT for TAVI Procedures
Acronym: CAVAREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Siemens Medical Solutions USA - CSG (Industry)
Responsible Party: Principal Investigator, Kenneth A. Fetterly, Ph.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-004257
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2016-01

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAVAREC images (Experimental): CAVAREC images from x-ray angiography
  Interventions: Other: CAVAREC Image Processing algorithm

INTERVENTIONS:
Other: CAVAREC Image Processing algorithm — After deployment of the TAVI prosthesis, other trans catheter valve, or stent, but before the patient care episode is completed, a set of rotational x-ray angiography images will be acquired and reconstructed using the clinical DyanCT and research CAVAREC algorithms.

SUMMARY:
The purpose of this work is to evaluate the feasibility of a new Cardiac Vascular Reconstruction (CAVAREC, Siemens Medical Systems, Germany) image reconstruction algorithm for use during transcatheter aortic valve implant (TAVI) procedures or interventional procedures to treat congenital or structural heart disease. CAVAREC utilizes the same x-ray projection images as currently acquired for clinical DynaCT. X-ray image acquisition to allow CAVAREC will occur during the interventional procedure after the TAVI device, other valve, or stent is implanted. If the participants already have a surgically-implanted TAVI device, stent or other device, and are having a cardiac catheterization, then an extra set of images will be acquired after your clinical care is complete, but before you leave the procedure room. The CAVAREC image processing algorithm will be implemented on an off-line workstation after the interventional procedure is complete. After the TAVI procedure, CAVAREC images will be quantitatively and qualitatively compared to Siemens DynaCT and cardiac CT images from Radiology. The results of this study will be used to direct further development of CAVAREC toward the end goal of providing improved imaging capabilities to guide TAVI, congenital heart, or structural heart treatment procedures.

DETAILED DESCRIPTION:
1. Compare utility of CAVAREC to standard DynaCT and cardiac CT for clinical assessment of the aortic valve and relevant, nearby anatomical structures.
2. Investigate the utility of CAVAREC to assess calcification within and surrounding the native aortic valve.
3. Investigate the utility of CAVAREC to assess procedural success, including prosthetic valve placement and annular anatomic correlates of paravalvular leak.
4. Validate utility of CAVAREC for images acquired during normal sinus rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Patients may either be scheduled for a TAVI procedure or scheduled for a cath lab appointment at any time after a TAVI procedure, or scheduled for device implant to treat congenital or structural heart disease.

Exclusion Criteria:

* Patient enrolled in research protocol with exclusions from simultaneous participation in another protocol
* Lack of research consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-02; Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Number of images of the aortic valve that are accurate | approx 2 hours after surgery
  Qualitative image assessment will be performed by Board Certified Cardiologists and/or Radiologists who are familiar with cardiac CT image manipulation and interpretation.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Fetterly, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States